CLINICAL TRIAL: NCT03153748
Title: New Therapeutic System of Ruptured Intracranial Aneurysms Based on Big Data From Chinese Population
Acronym: NATIONAL-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Qinghai Huang, Principal Investigator, Changhai Hospital
Other Study IDs: CHEC2017-074
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Treatment strategy
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at clarifying the current situation of Emergency treatment of aneurysmal subarachnoid hemorrhage (SAH) in China, and analyzing the safety and efficacy of the treatment strategy between interventional treatment and open surgery, so as to improve the diagnosis and treatment of aneurysmal SAH.

ELIGIBILITY:
Inclusion Criteria:

* patients presented with subarachnoid hemorrhage on CT or lumbar puncture.
* the intracranial hemorrhage was caused by rupture of aneurysm and was confirmed on CTA、MRA or DSA.
* patients willing to participate in this clinical trial and attach to regular follow up.

Exclusion Criteria:

* intracranial aneurysm correlating to AVM.
* dissection, false, traumatic and infectious aneurysms.
* the rupture of the aneurysm can not be confirmed on CTA、MRA or DSA.
* patients unwilling to participate in this clinical trial and attach to regular follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presented with subarachnoid hemorrhage and diagnosed with ruptured aneurysm at all age.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
mRS score | 1 year after treatment
  the mRS score after treatment
cure rate | 6 months after treatment
  the proportion of the cured-patient according Raymond Class

SECONDARY OUTCOMES:
recurrence rate | through study completion, an average of 1 year
  the proportion of the recurrence of the patient
complication rate | through study completion, an average of 1 year
  the proportion of complication happened after treatment including ischemic, hemorrhage, retreat, and so on

CONTACTS AND LOCATIONS:
Overall Officials: Qinghai Huang, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No